CLINICAL TRIAL: NCT02281773
Title: A Phase II Randomised, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Four Orally Administrated Doses of BI 409306 During a 12-week Treatment Period in Patients With Schizophrenia on Stable Antipsychotic Treatment
Brief Title: A Study to Investigate the Efficacy, Safety and Tolerability of Four Different Doses of BI 409306 Compared to Placebo Given for 12 Weeks in Patients With Schizophrenia on Stable Antipsychotic Treatment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.6; 2013-005015-28 (EudraCT Number)
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 409306

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- dose 1 (Experimental)
  Interventions: Drug: BI 409306 10 mg QD
- dose 2 (Experimental)
  Interventions: Drug: BI 498306 25 mg QD
- dose 3 (Experimental)
  Interventions: Drug: BI 498306 50 mg QD
- dose 4 (Experimental)
  Interventions: Drug: BI 409306 100 mg QD
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 409306 100 mg QD
  Arms: dose 4
Drug: BI 498306 50 mg QD
  Arms: dose 3
Drug: Placebo
  Arms: placebo
Drug: BI 498306 25 mg QD
  Arms: dose 2
Drug: BI 409306 10 mg QD
  Arms: dose 1

SUMMARY:
The objective of the study is to investigate the efficacy, safety and tolerability of four different doses of BI 409306 once daily compared to placebo given for 12 weeks in patients with schizophrenia on stable antipsychotic treatment.

ELIGIBILITY:
Inclusion criteria:

1. Patients with established diagnoses of schizophrenia (per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)) with the following clinical features:

   a) Clinically stable and are in the residual (non-acute) phase of their illness for at least 8 weeks b) Current antipsychotic and concomitant psychotropic medications must meet the criteria below: b)-1 Maintained on current atypical (second generation) antipsychotic medications (in any approved dosage form) other than Clozapine and on current dose for at least 8 weeks prior to randomisation, and/or b)-2 Maintained on current typical (first generation) antipsychotic medications and on current dose for at least 6 months, optionally combined with anticholinergics if treated with a stable dose for at least 6 months prior to randomisation, and/or b)-3 Maintained on current concomitant psychotropic medications other than anticholinergics, antiepileptics and lithium, and on current dose for at least 8 weeks prior to randomisation. Antiepileptics and lithium are allowed if initiated at least 6 months prior to randomisation.

   b)-4 Anticholinergics, antiepileptics and lithium have been washed out for at least 6 months prior to randomisation if the treatments that patients were using before entering the clinical trial are discontinued.

   c) Have no more than a "moderate" severity rating on hallucinations and delusions (Positive and Negative Syndrome Scale (PANSS)-positive syndrome Hallucinatory Behavior item score < =4 and Delusions item score < = 4) d) Have no more than a "moderate" severity rating on positive formal thought disorder (PANSS-positive syndrome Conceptual Disorganization item score < = 4) e) Have a minimal level of extrapyramidal symptoms (Simpson-Angus Scale total score < 6) and depressive symptoms (PANSS-general psychopathology syndrome Depression item score < = 4)
2. Male or female patients age 18 to 55 years
3. Patients must exhibit reliability, physiologic capability, and an educational level sufficient to comply with all protocol procedures,in the investigator's opinion.
4. Signed and dated written informed consent by date of Visit 1 in accordance with GCP and the local legislation. If the patient needs a legal representative, then this legal representative must give written informed consent as well.
5. Patients must have an identified informant who will be consistent throughout the study. The informant must interact with the subject at least 2 times a week.

Note: Informant ratings are needed for SCoRS global ratings at Randomisation Visit (Visit 2) and (early) End of Treatment Visit. In person informant ratings on the study visits are preferred whenever possible. However, if the informant is not available for in person ratings, telephone interview is acceptable. The informant must be available for a telephone interview at Visit 2 and (e)EOT Visit.

Exclusion criteria:

1. Patient treated with more than two antipsychotic medications (including more than two dosage forms)
2. Patient's cognitive impairment severity compromises the validity of the cognitive outcome measures, in the clinical judgment of the investigator
3. Any suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior)
4. Any suicidal ideation of type 4 or 5 in the Columbia Suicidal Severity Rating Scale (C-SSRS) in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
5. In the judgment of the investigator, any clinically significant finding of the medical examination (including BP, PR and ECG) or laboratory value deviating from normal or any evidence of a clinically significant concomitant disease or any other clinical condition that would jeopardize a patient's safety while participating in the clinical trial
6. History or diagnosis of symptomatic and unstable/uncontrolled gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hematological or hormonal disorders
7. For female patients:

   Pre-menopausal women (last menstruation < =1 year prior to informed consent) who:
   * are nursing or pregnant or
   * are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the trial until 28 days after the last treatment administration, and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, vasectomized partner, transdermal patch, intra uterine devices/systems (IUDs/IUSs), combined estrogen-progestin oral contraceptives as well as implantable or injectable hormonal contraceptives. Complete sexual abstinence (if acceptable by local health authorities) is allowed when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Double barrier methods are permissible (if acceptable by local health authorities, note that this is not an acceptable method in EU countries).

   For male patients:

   Men who are able to father a child, unwilling to be abstinent or use adequate contraception for the duration of study participation and for at least 28 days after treatment has ended.
8. Known history of HIV infection
9. Diseases of the central nervous system (including but not limited to any kind of seizures, stroke or any psychiatric disorders other than schizophrenia)
10. Any subject who on the Mini-international neuropsychiatric Interview (M.I.N.I.) has a categorical diagnosis of another current major psychiatric disorder.
11. History of malignancy within the last 5 years, except for basal cell carcinoma
12. Planned elective surgery requiring general anaesthesia, or hospitalisation for more than 1 day during the study period
13. Significant history of drug dependence or abuse (including alcohol, as defined in DSM-5-substance use disorder or in the opinion of the investigator) within the last two years prior to informed consent, or a positive urine drug screen for cocaine, opioid, PCP, amphetamine, heroin, or marijuana at screening
14. Patient needs to take long-acting hypnotics and anxiolytics (i.e. Diazepam)
15. Patients taking medications that are known to be strong or moderate CYP3A4 inhibitors
16. Participation in another trial with an investigational drug or procedure within 30 days or 6 half-lives (whichever is longer) or participation in another trial with any cognitive-enhancing therapy or procedure within 90 days prior to screening
17. Previous participation in any BI 409306 study
18. Not fluent in the language of the batteries/questionnaires which will be used in the country

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 518 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (43):
- United States (24):
  - K and S Professional Research Services, LLC, Little Rock, Arkansas
  - Comprehensive Clinical Development, Inc., Cerritos, California
  - Collaborative Neuroscience Network, Garden Grove, California
  - Pacific Institute of Medical Research, Los Angeles, California
  - SRSD, Inc. dba Synergy San Diego, National City, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Collaborative Neuroscience Network, Torrance, California
  - Comprehensive Clinical Development, Washington D.C., District of Columbia
  - Innovative Clinical Research, Lauderhill, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Atlanta Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Mid-America Clinical Research, LLC, St Louis, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Finger Lakes Research, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
- Canada (2):
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - Depression, Mood Disorders and Schizophrenia Treatment Centr, Burlington, Ontario
- Germany (3):
  - Universitätsklinikum Köln (AöR), Cologne
  - LVR-Klinikum Düsseldorf, Düsseldorf
  - Uniklinikum Heidelberg, Heidelberg
- Japan (10):
  - Fujita Health University Hospital, Aichi, Toyoake
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Kobe University Hospital, Hyogo, Kobe
  - Nara Medical University Hospital, Nara, Kashihara
  - Kansai Med. Univ. Med. Ctr., Osaka, Neuropsychiatry, Osaka, Moriguchi-city
  - Hizen Psychiatric Center, Saga, PSY, Saga, Kanzaki-gun
  - Iwaki Clinic, Tokushima, Psychosomatic Medicine, Tokushima, Anan
  - National Center Neurology and Psychiatry, Tokyo, Kodaira
  - Showa University Karasuyama Hospital, Tokyo, Setagaya
  - Showa University East Hospital, Tokyo, Shinagawa
- Taiwan (4):
  - Chang-Hua Christian Hospital, Changhua
  - Kai-Syuan Psychiatric Hospital, Kaohsiung City
  - NCKUH, Tainan
  - Taipei City Hospital, Taipei

REFERENCES:
- [Derived] Dorner-Ciossek C, Kroker KS, Rosenbrock H. Role of PDE9 in Cognition. Adv Neurobiol. 2017;17:231-254. doi: 10.1007/978-3-319-58811-7_9. PMID 28956335
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase II multi-centre, multi-national, randomised, double-blind, placebo-controlled parallel group trial to evaluate the efficacy, safety and tolerability of four orally administrated doses of BI 409306 during a 12-week treatment period in patients with schizophrenia on stable antipsychotic treatment.
Pre-assignment Details: Actually, 518 subjects were entered/randomised however 2 subjects were not treated and hence the number of subjects that started equals 516. One belongs to BI 409306 - 25 milligram and another to Placebo group.
Groups:
- BI 409306 - 10 Milligram: Subject received single oral dose of 10 milligram (mg) BI 409306 (film-coated tablet) along with two placebo matching 25mg/50mg tablets once daily for 12 weeks.
- BI 409306 - 25 Milligram: Subject received single oral dose of 25 milligram (mg) BI 409306 (film-coated tablet) along with placebo matching 10mg and 25mg/50mg tablet once daily for 12 weeks.
- BI 409306 - 50 Milligram: Subject received single oral dose of 50 milligram (mg) BI 409306 (film-coated tablet) along with placebo matching 10mg and 25mg/50mg tablet once daily for 12 weeks.
- BI 409306 - 100 Milligram: Subject received single oral dose of 100 milligram (mg) BI 409306 (2 film-coated tablets of 50 mg) along with placebo matching 10mg tablet once daily for 12 weeks.
- Placebo: Subject received single oral dose of placebo matching tablets (one placebo matching 10mg tablet and two placebo matching 25mg/50mg tablets) once daily for 12 weeks.
Period: Overall Study
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Started | 87 | 85 (Started are the treated patients) | 85 | 86 | 173 (Started are the treated patients)
Completed | 76 | 70 | 67 | 65 | 143
Not Completed | 11 | 15 | 18 | 21 | 30
Not completed — Adverse Event | 6 | 1 | 4 | 8 | 9
Not completed — Protocol Violation | 1 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 6 | 2 | 10
Not completed — Withdrawal by Subject | 2 | 8 | 6 | 6 | 8
Not completed — Other Reason | 0 | 4 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) was to consist of all patients who were randomised and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo | Total
Number analyzed (Participants) | 87 | 85 | 85 | 86 | 173 | 516
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (8.9) | 43.2 (9.4) | 41.4 (9.5) | 42.3 (9.5) | 41.5 (9.7) | 42.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 20 | 28 | 45 | 156
  Male | 53 | 56 | 65 | 58 | 128 | 360

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Composite Score of Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) After 12 Weeks of Treatment
Description: MCCB comprises 10 tests, which assess 7 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning problem solving, and social cognition. The composite score was calculated by summing over the standardised score of each domain for analysis and it varies from -20 to 99 with higher score indicating better outcome. The trial was set up as "learn and confirm" model including 2 stages. Stage 1 analysis was conducted to identify the meaningful cognition endpoint(s) (CANTAB domain(s)) and the selected endpoint(s) were to be pre-specified as the primary endpoint(s) for Stage 2 analysis. Since none of the CANTAB outcome measures was selected in the Stage 1 analysis at planned time based on the pre-specified criteria, the MCCB composite score was chosen as the primary endpoint in the Stage 2 analysis, as pre-defined.
Time Frame: Baseline and Week 12
Population: The full analysis set (FAS) was to consist of all randomisation patients who were treated with at least one dose of study drug and had a baseline and at least one post baseline on treatment primary endpoint MCCB composite score.
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 79 | 76 | 69 | 76 | 150
Unit on Scale | 1.2 (0.71) | 2.7 (0.74) | 2.8 (0.75) | 1.8 (0.73) | 2.5 (0.57)
Statistical Analysis 1: Comparison: BI 409306 - 10 Milligram vs Placebo; The restricted maximum likelihood (REML) based mixed effects model with repeated measurements (MMRM) was used with baseline value as fixed covariate and planned treatment, analysis visit, first test done, geographic region grouping 1, planned treatment by analysis visit and baseline value by analysis visit as fixed effects; Test type: Superiority or Other; p = 0.1256, Mixed Models Analysis — Due to the exploratory nature of this trial, no multiplicity adjustment was made. All statistical testing was performed using a two-sided, α=0.05 level of significance; Unstructured covariance structure has been used to fit the mixed model. Kenward-Roger was used to model degrees of freedom; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.76 to 0.34], Standard Error of Mean 0.79 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 10 mg minus Placebo
Statistical Analysis 2: Comparison: BI 409306 - 25 Milligram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7337, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.30 to 1.84], Standard Error of Mean 0.80 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 25 mg minus Placebo
Statistical Analysis 3: Comparison: BI 409306 - 50 Milligram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6994, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.31 to 1.95], Standard Error of Mean 0.83 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 50 mg minus Placebo
Statistical Analysis 4: Comparison: BI 409306 - 100 Milligram vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4270, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.19 to 0.93], Standard Error of Mean 0.79 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 100 mg minus Placebo

2. Primary Outcome: Occurrence of Serious Adverse Events (SAEs) (Including the Abnormalities of Physical Examination, Vital Signs, Electrocardiogram (ECG) Test and Laboratory Tests)
Description: Occurrence of serious adverse events (SAEs) (including the abnormalities of physical examination, vital signs, electrocardiogram (ECG) test and laboratory tests).
Time Frame: Up to 20 weeks
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 87 | 85 | 85 | 86 | 173
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 5.8

3. Primary Outcome: Occurrence of Protocol-specified Adverse Events of Special Interest (AESI)
Description: Occurrence of Protocol-specified adverse events of special interest (AESI).
Time Frame: Up to 20 weeks
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 87 | 85 | 85 | 86 | 173
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Dramatic Worsening of Disease State as Assessed by Positive and Negative Syndrome Scale (PANSS)
Description: Dramatic worsening of disease state as assessed by Positive and Negative Syndrome Scale (PANSS). It contains 30-items including seven positive symptom items, seven negative symptom items and 16 general psychopathology symptom items. Each item was scored on the same seven point severity scale. Fourteen of the PANSS items required input from an informant. Total score ranges from 30 to 210 (minimum is better). The descriptive statistics of change from baseline (CFB) in PANSS score at week 6 (W6) and week 12 (W12) are presented.
Time Frame: Baseline, Week 6 and Week 12
Population: TS
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 87 | 85 | 85 | 86 | 173
Unit on Scale
  W6-Number of participants analyzed:79,74,67,71,154 | -0.68 (6.022) | -0.28 (4.507) | -1.09 (5.415) | -1.20 (5.426) | -1.81 (5.895)
  W12-Number of participant analyzed:83,78,76,81,157 | -2.59 (5.342) | -0.97 (5.420) | -1.58 (6.990) | -0.94 (6.315) | -1.66 (6.942)

5. Primary Outcome: Suicidality as Assessed by Columbia Suicidal Severity Rating Scale (C-SSRS)
Description: C-SSRS: Number (%) of subjects with an event of Suicidal Ideation (Wish to be dead, Non-specific active suicidal thoughts, Active suicidal ideation with any methods (not plan) without intent to act, Active suicidal ideation with some intent to act without specific plan, Active suicidal ideation with specific plan and intent) or Suicidal Behavior (Preparatory acts or behavior, Aborted attempt, Interrupted attempt, Non-fatal suicide attempt, Completed suicide) or Self-injurious behavior without suicidal intent is presented. C-SSRS used only to evaluate whether the patient developed suicidal ideation or behavior and no composite score will be used. Questions in the 1st section of suicidal ideation and suicidal behavior assessments in C-SSRS are "yes" and "no" type questions. If patient had suicidal ideation or behavior, 2nd section will be performed to evaluate the details with the scale from 0 to 5 or 0 to 2 and the larger number means the more severe condition.
Time Frame: Up to 12 weeks
Population: TS (Number of subjects with a post baseline C-SSRS)
Measure: Number; unit: Percentage of Participants
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 84 | 84 | 79 | 85 | 166
Percentage of Participants | 0.0 (3.677) | 1.2 (3.262) | 2.5 (3.759) | 1.2 (3.497) | 3.6 (3.954)

6. Secondary Outcome: Change From Baseline in Everyday Functional Capacity as Measured by Schizophrenia Cognition Rating Scale (SCoRS) Global Ratings After 12 Weeks of Treatment
Description: Change from baseline in everyday functional capacity as measured by Schizophrenia Cognition Rating Scale (SCoRS) global ratings after 12 weeks of treatment. SCoRS is a 20-item interview-based assessment of cognitive deficits and the degree to which they affect day-to-day functions. Each item was rated on a 4-point scale. Higher ratings reflected a greater degree of impairment. The SCoRS global total scores is the sum of the 20 items and it varies from 20 to 80 with 20 being the best outcome and 80 being the worst. If any individual item was missing, it was imputed with the average of that patient's non missing responses. If >5 items were missing, the total score was missing.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 82 | 75 | 73 | 80 | 156
Unit on Scale | -2.2 (0.53) | -3.1 (0.56) | -2.0 (0.56) | -2.3 (0.54) | -2.5 (0.39)
Statistical Analysis 1: Comparison: BI 409306 - 10 Milligram vs Placebo; Analyses of covariance (ANCOVA) were used to assess between-group differences (BI 409306 group minus placebo group) in the modelled changes from baseline to Week 12. The dependent variable was the change from the baseline score at Week 12 during the treatment period adjusted for fixed categorical covariates of treatment as well as fixed continuous covariates of baseline score; Test type: Superiority or Other; p = 0.5972, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.9 to 1.6], Standard Error of Mean 0.66 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 10 mg minus Placebo
Statistical Analysis 2: Comparison: BI 409306 - 25 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3817, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.9 to 0.7], Standard Error of Mean 0.68 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 25 mg minus Placebo
Statistical Analysis 3: Comparison: BI 409306 - 50 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.4800, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.9 to 1.8], Standard Error of Mean 0.68 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 50 mg minus Placebo
Statistical Analysis 4: Comparison: BI 409306 - 100 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.7507, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.1 to 1.5], Standard Error of Mean 0.66 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 100 mg minus Placebo

7. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Scale Score After 12 Weeks of Treatment
Description: Change from baseline in Clinical Global Impressions-Severity (CGI-S) scale score after 12 weeks of treatment. The CGI-S is a one-item evaluation completed by the clinician on the patient's severity of psychopathology. The CGI-S was rated ordinally from one to 7. Higher scores indicate more severe symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 82 | 77 | 73 | 81 | 157
Unit on Scale | -0.1 (0.05) | -0.1 (0.05) | -0.1 (0.05) | -0.1 (0.05) | -0.1 (0.03)
Statistical Analysis 1: Comparison: BI 409306 - 10 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.9399, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 10 mg minus Placebo
Statistical Analysis 2: Comparison: BI 409306 - 25 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.9919, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.06 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 25 mg minus Placebo
Statistical Analysis 3: Comparison: BI 409306 - 50 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3027, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.06 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 50 mg minus Placebo
Statistical Analysis 4: Comparison: BI 409306 - 100 Milligram vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3901, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.06 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as BI 409306 100 mg minus Placebo

8. Secondary Outcome: Patient Global Impressions-Improvement (PGI-I) Scale Score Measured After 12 Weeks of Treatment
Description: Patient Global Impressions-Improvement (PGI-I) scale score measured after 12 weeks of treatment. The PGI of improvement is a simple evaluation completed by the patient to assess the patient's overall evaluation of his/her status. The PGI of improvement was rated ordinally from one to 7. Higher scores indicate more severe symptoms.
Time Frame: Up to 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 82 | 77 | 73 | 82 | 157
Unit on Scale | 2.988 (1.117) | 2.883 (1.124) | 3.192 (1.101) | 3.049 (1.342) | 3.038 (1.109)

9. Secondary Outcome: Change From Baseline in PANSS Negative Symptom Factor Score After 12 Weeks of Treatment (for Subset of Patients Diagnosed With Negative Symptom)
Description: Change from baseline in PANSS negative symptom factor score after 12 weeks of treatment (for subset of patients diagnosed with negative symptom). This outcome measure was not analysed due to low number of patients in the PANSS negative symptom subgroup. The PANSS negative symptom scale has 7 items. Each was rated from one to 7 points. The total factor score was the summation of the 7 points for each item, leading the total score ranging from 7 to 49.
Time Frame: Baseline and Week 12
Population: This endpoint was not analysed because as per internal Boehringer Ingelheim rules, descriptive statistics are not calculated if data is available for less than 2/3rds of participants.
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change in Psychopathology Symptoms as Assessed by Positive and Negative Syndrome Scale (PANSS)
Description: Change in psychopathology symptoms as assessed by Positive and Negative Syndrome Scale (PANSS). It contains 30-items including seven positive symptom items, seven negative symptom items and 16 general psychopathology symptom items. Each item was scored on the same seven point severity scale. Fourteen of the PANSS items required input from an informant. Total score ranges from 30 to 210 (minimum is better). The descriptive statistics of change from baseline (CFB) in PANSS score at week 6 (W6) and week 12 (W12) are presented.
Time Frame: Baseline, Week 6 and Week 12
Population: TS
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Number analyzed (Participants) | 87 | 85 | 85 | 86 | 173
Unit on Scale
  W6-Number of participants analyzed:79,74,67,71,154 | -0.39 (3.677) | -0.22 (3.262) | -0.31 (3.759) | -0.79 (3.497) | -0.99 (3.954)
  W12-Number of participant analyzed:83,78,76,81,157 | -1.36 (3.039) | -0.79 (3.277) | -0.68 (4.253) | -0.38 (3.587) | -0.76 (4.007)

ADVERSE EVENTS:
Time Frame: From first drug administration until 4 weeks after the last drug administration, up to 16 weeks
Arm/Group | BI 409306 - 10 Milligram | BI 409306 - 25 Milligram | BI 409306 - 50 Milligram | BI 409306 - 100 Milligram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/85 | 0/85 | 0/86 | 10/173
Other Adverse Events (participants affected / at risk) | 5/87 | 9/85 | 9/85 | 12/86 | 12/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 - 10 Milligram (N=87) | BI 409306 - 25 Milligram (N=85) | BI 409306 - 50 Milligram (N=85) | BI 409306 - 100 Milligram (N=86) | Placebo (N=173)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 - 10 Milligram (N=87) | BI 409306 - 25 Milligram (N=85) | BI 409306 - 50 Milligram (N=85) | BI 409306 - 100 Milligram (N=86) | Placebo (N=173)
Photophobia (Eye disorders) | 0 | 2 | 2 | 6 | 2
Visual brightness (Eye disorders) | 0 | 2 | 3 | 6 | 0
Headache (Nervous system disorders) | 5 | 5 | 4 | 1 | 10

LIMITATIONS AND CAVEATS:
"Change from baseline in PANSS negative symptom factor score after 12 weeks of treatment" was not analysed because as per internal BI rules, descriptive statistics are not calculated if data is available for less than 2/3rds of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.